CLINICAL TRIAL: NCT04189367
Title: A Prospective Study on the Treatment of Burning Mouth Syndrome With Integration of Traditional Chinese Medicine(TCM) and Western Medicine Based on TCM Syndrome Differentiation
Brief Title: Treatment of Burning Mouth Syndrome With Integration of Traditional Chinese Medicine and Western Medicine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, MENG LING CHIANG, DDS, Director, Head of Oral Pathology and Oral Diagnosis, Principal Investigator, Assistant Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201802359A3C601; NMRPG3J6101 (Other Grant/Funding Number: Ministry of Science and Technology, Taiwan)
Record Dates: First submitted 2019-12-03; First posted 2019-12-06 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Burning Mouth Syndrome
Keywords: Burning Mouth Syndrome; Traditional Chinese Medicine; Automatic Tongue Diagnosis System; Body Constitution Questionnaire
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Western medicine + TCM (Experimental): 1. Meet the conditions of inclusion and exclusion, seek the consent of the patient, and fill out the informed consent.
  2. Blood test and physiological assessment, and do the TCM model.
  3. Primary type BMS patients receive clonazepam 0.5 mg PO every day before sleep or twice a day for 12 weeks
  4. Secondary BMS patients receive nutritional supplements according to the patient's hematic deficiency status for 12 weeks.
  5. TCM therapy: one bag of "Qingre Liangkou Ningxin Fang", three times a day for 12 weeks.
  Interventions: Drug: Traditional Chinese Medicine; Drug: Western medicine
- Western medicine (Active Comparator): 1. Meet the conditions of inclusion and exclusion, seek the consent of the patient, and fill out the informed consent.
  2. Blood test and physiological assessment, and do the TCM model.
  3. Primary type BMS patients receive clonazepam 0.5 mg PO every day before sleep or twice a day for 12 weeks
  4. Secondary BMS patients receive nutritional supplements according to the patient's hematic deficiency status for 12 weeks.
  Interventions: Drug: Western medicine

INTERVENTIONS:
Drug: Traditional Chinese Medicine — One bag of " Qingre Liangkou Ningxin Fang" at a time, three times a day for 12 weeks.
  Other Names: TCM
  Arms: Western medicine + TCM
Drug: Western medicine — Western medicine includes:
  1. clonazepam 0.5mg every day before sleep or twice a day for 12 weeks
  2. Nutritional supplement: vitamin B12, folic acid, iron, zinc, vitamin B complex depending on the hematic deficiency, for 12 weeks
  Other Names: WM

SUMMARY:
This study is an open-label randomized controlled trial of the efficacy of the integration of Traditional Chinese medicine (TCM) and western medicine based on TCM syndrome differentiation. The hypothesis is (1) TCM model can identify the primary and secondary type burning mouth syndrome (BMS); (2) TCM model can identify BMS after treatment with western medicine; (3) There is a positive effect of TCM in treating BMS.

DETAILED DESCRIPTION:
BMS patients will be classified into the primary type and secondary type according to the patients' clinical histories and laboratory examinations. The secondary BMS only includes nutritional deficiency, such as Vitamin B12, folate, iron, zinc. At first, the primary BMS patients are treated with 0.5~1 mg clonazepam every day before sleep for 8 weeks. The secondary BMS patients are treated with vitamin B12, folate, iron and zinc according to the patient's nutritional deficiency status. Patients with no improvement or little improvement after the first stage of Western medicine management will be arranged to receive traditional Chinese medicine (TCM) therapy. All patients will receive the TCM model, including TCM doctor, automatic tongue diagnostic system (ATDS), and body constitutional questionnaire (BCQ), evaluations.

The results of this study are expected to understand whether adjuvant TCM treatment of BMS can improve treatment efficacy. The investigators will understand whether the constitution pattern may be a predictive indicator of efficacy for western BMS. The investigators will find a diagnostic indicator for the TCM model and apply it to the assessment of the prognosis of BMS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who signed the informed consent
2. The clinical diagnosis was primary or secondary type BMS patient
3. ≥ 20-year-old
4. Female
5. Willing to take Traditional Chinese Medicine

Exclusion Criteria:

1. History of an angiotensin-converting enzyme inhibitor (ACEI) taking
2. Autoimmune disease
3. Poor kidney function
4. Unwilling to take Traditional Chinese Medicine
5. Male
6. Participants who have been treated with TCM or Acupuncture within a month
7. Participants who have been treated with medicine for burning mouth syndrome

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility is based on the different prescriptions of Traditional Chinese Medicine for female and male subjects, not on self-representation of gender identity.
Enrollment: 80 (Estimated)
Dates: Start 2020-06-20 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Global perceived effect (GPE) | after treatment 1 week, 3 weeks, 6 weeks, 9weeks, 12weeks
  GPE is defined as symptoms improvement change compared to baseline, 1=worse; 2=no difference; 3=mild improvement; 4=much improvement; 5=totally improvement.
  The responder is defined to be the subject occurring at least one of the defined effective events: (1) GPE ≥2 after treatment for burning sensation; (2) GPE ≥2 after treatment for sleep; (3) GPE ≥2 after treatment for dry mouth; (4) GPE ≥2 after treatment for taste change. (5) GPE ≥2 after treatment for her other uncomfortable.
Numerical Rating Scale (NRS) | baseline, after treatment 1 week, 3 weeks, 6 weeks, 9weeks, 12weeks
  NRS is defined as 0=no pain, scale from 1 to 10 (mild to very severe).
  The responder is defined to be the subject occurring at least one of the defined effective events: (1) NRS ≤ 1 after treatment; (2) NRS change from baseline ≥ 50% after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Ling Chiang, DDS,MS, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grushka M, Epstein JB, Gorsky M. Burning mouth syndrome. Am Fam Physician. 2002 Feb 15;65(4):615-20. PMID 11871678
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Background] Jaaskelainen SK. Is burning mouth syndrome a neuropathic pain condition? Pain. 2018 Mar;159(3):610-613. doi: 10.1097/j.pain.0000000000001090. PMID 29257770
- [Background] Liu YF, Kim Y, Yoo T, Han P, Inman JC. Burning mouth syndrome: a systematic review of treatments. Oral Dis. 2018 Apr;24(3):325-334. doi: 10.1111/odi.12660. Epub 2017 Mar 30. PMID 28247977
- [Background] McMillan R, Forssell H, Buchanan JA, Glenny AM, Weldon JC, Zakrzewska JM. Interventions for treating burning mouth syndrome. Cochrane Database Syst Rev. 2016 Nov 18;11(11):CD002779. doi: 10.1002/14651858.CD002779.pub3. PMID 27855478
- [Background] Minguez-Sanz MP, Salort-Llorca C, Silvestre-Donat FJ. Etiology of burning mouth syndrome: a review and update. Med Oral Patol Oral Cir Bucal. 2011 Mar 1;16(2):e144-8. doi: 10.4317/medoral.16.e144. PMID 21217613
- [Background] Zakrzewska JM, Forssell H, Glenny AM. Interventions for the treatment of burning mouth syndrome. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD002779. doi: 10.1002/14651858.CD002779.pub2. PMID 15674897
- [Result] Adamo D, Sardella A, Varoni E, Lajolo C, Biasotto M, Ottaviani G, Vescovi P, Simonazzi T, Pentenero M, Ardore M, Spadari F, Bombeccari G, Montebugnoli L, Gissi DB, Campisi G, Panzarella V, Carbone M, Valpreda L, Giuliani M, Aria M, Lo Muzio L, Mignogna MD. The association between burning mouth syndrome and sleep disturbance: A case-control multicentre study. Oral Dis. 2018 May;24(4):638-649. doi: 10.1111/odi.12807. Epub 2018 Mar 13. PMID 29156085
- [Result] Cavalcanti DR, da Silveira FR. Alpha lipoic acid in burning mouth syndrome--a randomized double-blind placebo-controlled trial. J Oral Pathol Med. 2009 Mar;38(3):254-61. doi: 10.1111/j.1600-0714.2008.00735.x. Epub 2009 Jan 23. PMID 19175713
- [Result] Chang CM, Wu PC, Chiang JH, Wei YH, Chen FP, Chen TJ, Pan TL, Yen HR, Chang HH. Integrative therapy decreases the risk of lupus nephritis in patients with systemic lupus erythematosus: A population-based retrospective cohort study. J Ethnopharmacol. 2017 Jan 20;196:201-212. doi: 10.1016/j.jep.2016.12.016. Epub 2016 Dec 12. PMID 27974236
- [Result] Chang YY, Tsai YT, Lai JN, Yeh CH, Lin SK. The traditional Chinese medicine prescription patterns for migraine patients in Taiwan: a population-based study. J Ethnopharmacol. 2014 Feb 12;151(3):1209-1217. doi: 10.1016/j.jep.2013.12.040. Epub 2014 Jan 2. PMID 24389028
- [Result] Chen HY, Lin YH, Wu JC, Chen YC, Yang SH, Chen JL, Chen TJ. Prescription patterns of Chinese herbal products for menopausal syndrome: analysis of a nationwide prescription database. J Ethnopharmacol. 2011 Oct 11;137(3):1261-6. doi: 10.1016/j.jep.2011.07.053. Epub 2011 Aug 2. PMID 21824510
- [Result] Chen HY, Huang BS, Lin YH, Su IH, Yang SH, Chen JL, Huang JW, Chen YC. Identifying Chinese herbal medicine for premenstrual syndrome: implications from a nationwide database. BMC Complement Altern Med. 2014 Jun 27;14:206. doi: 10.1186/1472-6882-14-206. PMID 24969368
- [Result] Chen LL, Lin JS, Lin JD, Chang CH, Kuo HW, Liang WM, Su YC. BCQ+: a body constitution questionnaire to assess Yang-Xu. Part II: Evaluation of reliability and validity. Forsch Komplementmed. 2009 Feb;16(1):20-7. doi: 10.1159/000197770. Epub 2009 Feb 17. PMID 19295226
- [Result] Chen YL, Lee CY, Huang KH, Kuan YH, Chen M. Prescription patterns of Chinese herbal products for patients with sleep disorder and major depressive disorder in Taiwan. J Ethnopharmacol. 2015 Aug 2;171:307-16. doi: 10.1016/j.jep.2015.05.045. Epub 2015 Jun 9. PMID 26068429
- [Result] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Result] Femiano F, Gombos F, Scully C, Busciolano M, De Luca P. Burning mouth syndrome (BMS): controlled open trial of the efficacy of alpha-lipoic acid (thioctic acid) on symptomatology. Oral Dis. 2000 Sep;6(5):274-7. doi: 10.1111/j.1601-0825.2000.tb00138.x. PMID 11002408
- [Result] Grushka M, Epstein J, Mott A. An open-label, dose escalation pilot study of the effect of clonazepam in burning mouth syndrome. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1998 Nov;86(5):557-61. doi: 10.1016/s1079-2104(98)90345-6. PMID 9830647
- [Result] Heckmann SM, Kirchner E, Grushka M, Wichmann MG, Hummel T. A double-blind study on clonazepam in patients with burning mouth syndrome. Laryngoscope. 2012 Apr;122(4):813-6. doi: 10.1002/lary.22490. Epub 2012 Feb 16. PMID 22344742
- [Result] Hens MJ, Alonso-Ferreira V, Villaverde-Hueso A, Abaitua I, Posada de la Paz M. Cost-effectiveness analysis of burning mouth syndrome therapy. Community Dent Oral Epidemiol. 2012 Apr;40(2):185-92. doi: 10.1111/j.1600-0528.2011.00645.x. Epub 2011 Nov 1. PMID 22044166
- [Result] Hidaka T, Yonezawa R, Saito S. Kami-shoyo-san, Kampo (Japanese traditional medicine), is effective for climacteric syndrome, especially in hormone-replacement-therapy-resistant patients who strongly complain of psychological symptoms. J Obstet Gynaecol Res. 2013 Jan;39(1):223-8. doi: 10.1111/j.1447-0756.2012.01936.x. Epub 2012 Jul 6. PMID 22765925
- [Result] Hsu PC, Tsai YT, Lai JN, Wu CT, Lin SK, Huang CY. Integrating traditional Chinese medicine healthcare into diabetes care by reducing the risk of developing kidney failure among type 2 diabetic patients: a population-based case control study. J Ethnopharmacol. 2014 Oct 28;156:358-64. doi: 10.1016/j.jep.2014.08.029. Epub 2014 Aug 29. PMID 25178949
- [Result] Imura H, Shimada M, Yamazaki Y, Sugimoto K. Characteristic changes of saliva and taste in burning mouth syndrome patients. J Oral Pathol Med. 2016 Mar;45(3):231-6. doi: 10.1111/jop.12350. Epub 2015 Aug 21. PMID 26293497
- [Result] Kuten-Shorrer M, Treister NS, Stock S, Kelley JM, Ji YD, Woo SB, Lerman MA, Palmason S, Sonis ST, Villa A. Safety and tolerability of topical clonazepam solution for management of oral dysesthesia. Oral Surg Oral Med Oral Pathol Oral Radiol. 2017 Aug;124(2):146-151. doi: 10.1016/j.oooo.2017.05.470. Epub 2017 May 11. PMID 28606830
- [Result] Lien AS, Jiang YD, Mou CH, Sun MF, Gau BS, Yen HR. Integrative traditional Chinese medicine therapy reduces the risk of diabetic ketoacidosis in patients with type 1 diabetes mellitus. J Ethnopharmacol. 2016 Sep 15;191:324-330. doi: 10.1016/j.jep.2016.06.051. Epub 2016 Jun 20. PMID 27340102
- [Result] Lee AL, Chen BC, Mou CH, Sun MF, Yen HR. Association of Traditional Chinese Medicine Therapy and the Risk of Vascular Complications in Patients With Type II Diabetes Mellitus: A Nationwide, Retrospective, Taiwanese-Registry, Cohort Study. Medicine (Baltimore). 2016 Jan;95(3):e2536. doi: 10.1097/MD.0000000000002536. PMID 26817897
- [Result] Lin JD, Chen LL, Lin JS, Chang CH, Huang YC, Su YC. BCQ-: a body constitution questionnaire to assess Yin-Xu. Part I: establishment of a provisional version through a Delphi process. Forsch Komplementmed. 2012;19(5):234-41. doi: 10.1159/000343580. Epub 2012 Oct 18. PMID 23128097
- [Result] Lin SK, Tsai YT, Lai JN, Wu CT. Demographic and medication characteristics of traditional Chinese medicine users among dementia patients in Taiwan: a nationwide database study. J Ethnopharmacol. 2015 Feb 23;161:108-15. doi: 10.1016/j.jep.2014.12.015. Epub 2014 Dec 17. PMID 25527314
- [Result] Lin YC, Chang TT, Chen HJ, Wang CH, Sun MF, Yen HR. Characteristics of traditional Chinese medicine usage in children with precocious puberty: A nationwide population-based study. J Ethnopharmacol. 2017 Jun 9;205:231-239. doi: 10.1016/j.jep.2017.05.006. Epub 2017 May 10. PMID 28499829
- [Result] Lin YR, Wu MY, Chiang JH, Yen HR, Yang ST. The utilization of traditional Chinese medicine in patients with dysfunctional uterine bleeding in Taiwan: a nationwide population-based study. BMC Complement Altern Med. 2017 Aug 29;17(1):427. doi: 10.1186/s12906-017-1939-1. PMID 28851349
- [Result] Lo LC, Chen YF, Chen WJ, Cheng TL, Chiang JY. The Study on the Agreement between Automatic Tongue Diagnosis System and Traditional Chinese Medicine Practitioners. Evid Based Complement Alternat Med. 2012;2012:505063. doi: 10.1155/2012/505063. Epub 2012 Aug 8. PMID 22924055
- [Result] Lo LC, Cheng TL, Chiang JY, Damdinsuren N. Breast cancer index: a perspective on tongue diagnosis in traditional chinese medicine. J Tradit Complement Med. 2013 Jul;3(3):194-203. doi: 10.4103/2225-4110.114901. PMID 24716178
- [Result] Lo LC, Cheng TL, Chen YJ, Natsagdorj S, Chiang JY. TCM tongue diagnosis index of early-stage breast cancer. Complement Ther Med. 2015 Oct;23(5):705-13. doi: 10.1016/j.ctim.2015.07.001. Epub 2015 Jul 10. PMID 26365451
- [Result] Ma YC, Lin CC, Li CI, Chiang JH, Li TC, Lin JG. Traditional Chinese medicine therapy improves the survival of systemic lupus erythematosus patients. Semin Arthritis Rheum. 2016 Apr;45(5):596-603. doi: 10.1016/j.semarthrit.2015.09.006. PMID 26522135
- [Result] Park DM, Kim SH, Park YC, Kang WC, Lee SR, Jung IC. The comparative clinical study of efficacy of Gamisoyo-San (Jiaweixiaoyaosan) on generalized anxiety disorder according to differently manufactured preparations: multicenter, randomized, double blind, placebo controlled trial. J Ethnopharmacol. 2014 Dec 2;158 Pt A:11-7. doi: 10.1016/j.jep.2014.10.024. Epub 2014 Oct 23. PMID 25456420
- [Result] Pinder RM, Brogden RN, Speight TM, Avery GS. Clonazepam: a review of its pharmacological properties and therapeutic efficacy in epilepsy. Drugs. 1976 Nov;12(5):321-61. doi: 10.2165/00003495-197612050-00001. PMID 976134
- [Result] Puhakka A, Forssell H, Soinila S, Virtanen A, Roytta M, Laine M, Tenovuo O, Teerijoki-Oksa T, Jaaskelainen SK. Peripheral nervous system involvement in primary burning mouth syndrome--results of a pilot study. Oral Dis. 2016 May;22(4):338-44. doi: 10.1111/odi.12454. Epub 2016 Feb 26. PMID 26847146
- [Result] Qu Y, Gan HQ, Mei QB, Liu L. Study on the effect of Jia-Wei-Xiao-Yao-San decoction on patients with functional dyspepsia. Phytother Res. 2010 Feb;24(2):245-8. doi: 10.1002/ptr.2920. PMID 19610028
- [Result] Sun A, Lin HP, Wang YP, Chen HM, Cheng SJ, Chiang CP. Significant reduction of serum homocysteine level and oral symptoms after different vitamin-supplement treatments in patients with burning mouth syndrome. J Oral Pathol Med. 2013 Jul;42(6):474-9. doi: 10.1111/jop.12043. Epub 2013 Jan 9. PMID 23297780
- [Result] Sikora M, Verzak Z, Matijevic M, Vcev A, Siber S, Music L, Carek A. Anxiety and Depression Scores in Patients with Burning Mouth Syndrome. Psychiatr Danub. 2018 Dec;30(4):466-470. doi: 10.24869/psyd.2018.466. PMID 30439807
- [Result] Su YC, Chen LL, Lin JD, Lin JS, Huang YC, Lai JS. BCQ+: a body constitution questionnaire to assess Yang-Xu. Part I: establishment of a first final version through a Delphi process. Forsch Komplementmed. 2008 Dec;15(6):327-34. doi: 10.1159/000175938. Epub 2008 Dec 5. PMID 19142042
- [Result] Terauchi M, Hiramitsu S, Akiyoshi M, Owa Y, Kato K, Obayashi S, Matsushima E, Kubota T. Effects of three Kampo formulae: Tokishakuyakusan (TJ-23), Kamishoyosan (TJ-24), and Keishibukuryogan (TJ-25) on Japanese peri- and postmenopausal women with sleep disturbances. Arch Gynecol Obstet. 2011 Oct;284(4):913-21. doi: 10.1007/s00404-010-1779-4. Epub 2010 Dec 1. PMID 21120510
- [Result] Tsai DS, Chang YS, Li TC, Peng WH. Prescription pattern of Chinese herbal products for hypertension in Taiwan: a population-based study. J Ethnopharmacol. 2014 Sep 29;155(3):1534-40. doi: 10.1016/j.jep.2014.07.047. Epub 2014 Aug 1. PMID 25091464
- [Result] Yang YH, Chen PC, Wang JD, Lee CH, Lai JN. Prescription pattern of traditional Chinese medicine for climacteric women in Taiwan. Climacteric. 2009 Dec;12(6):541-7. doi: 10.3109/13697130903060081. PMID 19905906
- [Result] Yu MC, Lin SK, Lai JN, Wei JC, Cheng CY. The traditional Chinese medicine prescription patterns of Sjogren׳s patients in Taiwan: a population-based study. J Ethnopharmacol. 2014 Aug 8;155(1):435-42. doi: 10.1016/j.jep.2014.05.049. Epub 2014 Jun 4. PMID 24905866